CLINICAL TRIAL: NCT06271174
Title: Impact Evaluation of Perioperative Locoregional Analgesia on Persistent Postoperative Pain in Children After Orthopedic Surgery for Traumatology : a Prospective, Single Center, Randomised Controlled Study.
Brief Title: Avoid With Locoregional Analgesia Persistant Postoperative Pain In Children
Acronym: AWA3PASIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC23_0009
Record Dates: First submitted 2023-07-19; First posted 2024-02-21 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Persistent Postoperative Pain
Keywords: Persistent Postoperative Pain; Post-surgical chronic pain; Children; Loco-regional Analgesia; Orthopedic surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Mepivacaine; Anesthetics, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loco-Regional Analgesia (Experimental): Patients will receive Loco-Regional Analgesia during General Anesthesia, and systemic analgesia if necessary
  * Carbocaine
  Interventions: Drug: Carbocaine; Drug: Profofol and/or Suxaméthonium and/or Sévoflurane
- Systemic Analgesia Only (Active Comparator): Patients will just receive General Anesthesia and systemic analgesia.
  _ Profofol and/or Suxaméthonium and/or Sévoflurane
  Interventions: Drug: Profofol and/or Suxaméthonium and/or Sévoflurane

INTERVENTIONS:
Drug: Carbocaine — After general anesthesia and before incision, patients will receive loco-regional analgesia.
  Carbocaïne will be injected around the nerve responsible of the innervation of the operated area by echography guidance.
  Other Names: Loco regional Analgesia
  Arms: Loco-Regional Analgesia
Drug: Profofol and/or Suxaméthonium and/or Sévoflurane — General anesthesia
  Anesthetic induction is performed on a full stomach using :
  * Intravenous hypnotic Propofol 2-5 mg/kg
  * A rapid-acting intravenous curare Suxamethonium 1 mg/kg
  On an empty stomach :
  - An intravenous hypnotic Propofol 2 to 5 mg/kg or/and an inhalatory hypnotic, Sevoflurane, as anesthetic co-induction by these 2 agents is generally used in pediatrics.
  Other Names: General anesthetic

SUMMARY:
Persistent postoperative pain is a substantial pain (scores 4-10 using a 0-10 numeric scale) that develops 3 months after surgery.

Persistent postoperative pain can be a problem even in ambulatory surgery. Loco-regional analgesia could prevent the occurrence of this pathology but contradictory results are found in ancient studies.

This study is the first randomized controlled study in children about loco-regional analgesia and persistent postoperative pain in traumatologic orthopedic surgery.

One interventional arm will receive a locoregional analgesia after general anesthesia and before incision. The other arm will only receive systemic analgesia during general anesthesia.

The incidence of persistent postoperative pain at 3, 6 and 12 months will be compared in these two groups.

The goal is to show the decrease of the incidence of the persistent postoperative pain in the group "locoregional analgesia".

DETAILED DESCRIPTION:
Patients between 5 years old and 15 years, 3 months old operated for a traumatologic orthopedic surgery in CHU Nantes will be included in this study.

Patients between 5 years old and 15 years, 3 months old operated for a traumatologic orthopedic surgery in CHU Nantes will be included in this study.

They will be randomized in two groups. General anesthesia will be administered in both groups.

One arm will receive a locoregional analgesia guiding by echography before incision with a local anesthetic (Carbocaïne) and a systemic analgesia if necessary. One arm will only receive a systemic analgesia.

The drugs used for general anesthesia and systemic analgesia will be standardized in the two groups.

The incidence of persistent postoperative pain at 3, 6 and 12 months will be compared in both arms. A screening of a neuropathic pain will be realized if a pain exists.

The consumption of opioids the first 24 postoperative hours, the time spent in the post interventional care unit and the incidence of nausea, vomiting will also be compared.

The goal is to show the decrease of the incidence of the persistent postoperative pain and a better recovery in the post interventional care unit in the group "locoregional analgesia".

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 years old and 15 years and 3 months
* Traumatologic orthopedic surgery in CHU Nantes
* Conscious patient (Glasgow score =15)
* Patients able to give a verbal assessment of their pain
* No contraindication to Locoregional Analgesia
* Patient member of the social security system
* Oral consent of the patient
* Signed consent of one of the two holders of parental authority

Exclusion Criteria:

* Refusal to participate of the patient or one of the two holders of parental authority
* Neurologic deficit of the operated limb before intervention
* Ischemia of the operated limb before intervention
* Polytraumatized patient
* Allergia to Carbocaïne
* Atrioventricular conduction disorders
* Patient included in an other study about analgesia
* Anticoagulant treatment
* Uncontrolled epilepsy despite treatment
* Porphyria

Ages: 5 Years to 183 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Persistent Postoperative Pain | 3 months after surgery
  Numerical Scale of pain superior to 3 (0 to 10). 0 : no pain - better outcome 10 : max of pain - worse outcome

SECONDARY OUTCOMES:
Screening of neuropathic pain if persistent postoperative pain - 3 months | 3 months after surgery.
  DN4 score (0 to 10) - Self-assessment scale for estimating the probability of neuropathic pain Patient score is equal to or greater than 4/10, the test is positive 0 : minimum value / better outcome 10 : maximul value / worse outcome
Screening of neuropathic pain if persistent postoperative pain - 6 months | 6 months after surgery.
  DN4 score (0 to 10) - Self-assessment scale for estimating the probability of neuropathic pain Patient score is equal to or greater than 4/10, the test is positive 0 : minimum value / better outcome 10 : maximul value / worse outcome
Screening of neuropathic pain if persistent postoperative pain - 12 months | 12 months after surgery.
  DN4 score (0 to ten) - Self-assessment scale for estimating the probability of neuropathic pain Patient score is equal to or greater than 4/10, the test is positive 0 : minimum value / better outcome 10 : maximul value / worse outcome
1st EN score in immediate post-operative ICU before morphine titration | in Post Interventional Care Unit after the surgery
  Numerical Scale of pain (0 to 10) 0 : no pain - better outcome 10 : max of pain - worse outcome
Persistent postoperative pain at 6 months. | 6 months after surgery.
  Numerical Scale of pain (0 to 10) 0 : no pain - better outcome 10 : max of pain - worse outcome
Persistent postoperative pain at 12 months. | 12 months after surgery.
  Numerical Scale of pain (0 to 10) 0 : no pain - better outcome 10 : max of pain - worse outcome
Postoperative nausea and vomiting | In Post Interventional Care Unit - after the surgery-
  presence or absence
Time in Post Interventional Care Unit | In Post Interventional Care Unit - after the surgery -
  Evaluation in minutes.
Opioïd dose received - Per-operative | Per-operative
  Evaluation in milligrammes
Opioïd dose received - in Post Interventional Care Unit | in Post Interventional Care Unit after the surgery-
  Evaluation in milligrammes
Opioïd dose received | during the first post-operative 24 hours in the surgery department
  Evaluation in milligrammes
Intravenous Morphine dose received in Post Interventional Care Unit | in Post Interventional Care Unit after the surgery-
  Evaluation in milligrammes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France